CLINICAL TRIAL: NCT06145334
Title: VOICES Socials for Older Veterans With Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D4894-P; 1I02RX004872-01P0 (Other Grant/Funding Number: RR&D)
Record Dates: First submitted 2023-11-14; First posted 2023-11-24 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Depression; Loneliness; Isolation
Keywords: Veteran; Depression; Loneliness; Isolation; Veteran Socials; Community; Socialization; Older Adults
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Twenty Veterans aged 65 or older with depression will engage in the intervention, Veterans Socials (VS). Veterans will receive 90-minutes of weekly social engagement in a community-setting in accordance with the VS manual. Each week will focus on social connections, engagement in social activities, and reinforcing behaviors that give individuals meaning and purpose. Each VS will be held in a community setting across 4 months. The investigators will evaluate the feasibility of VS including fidelity, retention, acceptability of the intervention and preliminary outcomes around social functioning.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Veterans Social (Experimental): Peer-led weekly community-based social groups (16 weeks)
  Interventions: Behavioral: Veterans Social

INTERVENTIONS:
Behavioral: Veterans Social — Peer-led weekly community-based social groups (16 weeks) that are current treatment at the study site.
  Other Names: VOICES Veterans Social

SUMMARY:
VOICES Veterans Socials (VS) support Veterans in the community through weekly social groups. Veterans socials have the potential to improve social functioning, mental health symptoms, and create lasting social support. This project aims to evaluate and improve Veterans Socials to help older Veterans with depression by adapting materials, interviewing VS attendees, and collecting questionnaires. The goal is to improve the program based on the results for future use and research.

DETAILED DESCRIPTION:
VOICES Veterans Socials is a peer-led weekly social group based in the community designed to promote sustainable social support among Veterans. The research seeks to adapt and conduct a preliminary evaluation of the Veterans Socials (VS) intervention with older Veterans. The study will develop a training procedure for VS facilitators and evaluate an open trial of this intervention. This study will determine whether a larger-scale, more definitive VS study is indicated

Phase 1: 13 total participants will engage in semi-structured interviews about barriers to social engagement, challenges around community-based activities, social support acquisition, and how their age and Veteran status intersects with these constructs.

Phase 2: 20 participants will be recruited for VOICES Veterans Socials (VS) which will be conducted in 2-4 community-based social groups, with 5-10 participants in each social group. The investigators will conduct data collection on three occasions; at enrollment (pre; 0 months), at intervention completion (post; including semi-structured interview; 4 months) and at follow-up (7 months).

VS Procedures. Twenty Veterans aged 65 or older with depression will engage in VS. Veterans will receive 90-minutes of weekly social engagement in a community-setting in accordance with the VS manual. Each week will focus on social connections, engagement in social activities, and reinforcing behaviors that give individuals meaning and purpose.

ELIGIBILITY:
Inclusion Criteria:

* Documented depressive disorder or score of 2 or more on the Patient Health Questionnaire-2 (PHQ-2)
* Capacity to consent as determined by the University of California, San Diego Brief Assessment of Capacity to Consent (UBACC)
* Score of 1 or more on question 3 of the UCLA-3 OR score of 3 or less on question 4 of the Lubben Social Network Scale 6 (LSNS-6)

Exclusion Criteria:

* DSM-5 diagnosis of Schizophrenia Spectrum Disorder or Bipolar Disorder
* Symptoms of psychosis that would interfere with study participation
* Probable Dementia as determined by the 6-item Cognitive Impairment Screener
* Suicidal ideation with plan or intent
* Non-English speaking
* Active substance use disorder (DSM-5) (within 30 days of study entry)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 19 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2026-01-01 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire -2 (PHQ-2)- CHANGE IS BEING ASSESSED | Baseline, 4 month, 7 month
  Patient Health Questionnaire -2 (PHQ-2) is a 2-item screening tool that includes the first two items of the PHQ-9. It is frequently used to identify patients in which major depressive disorder is likely. A PHQ-2 score ranges from 0-6, with a score of 3 or greater indicating major depressive disorder is likely.
Beck Depression Inventory-II (BDI-II)- CHANGE IS BEING ASSESSED | Baseline, 4 month, 7 month
  Beck Depression Inventory-II (BDI-II) is a 21-item self-administered screening tool measuring the severity of depression in adolescents and adults. Higher scores indicate more depressive symptoms. The highest score is 63 and the lowest possible score for the test is zero.
Duke Social Support Index (DSSI)- CHANGE IS BEING ASSESSED | Baseline, 4 month, 7 month
  The Duke Social Support Index (DSSI) includes twenty-three items in three subscales: social interaction, subjective social support, and instrumental support). They are scored using a 3-point Likert scale and together assess social isolation. The scale ranges from 7 to 21 with higher scores indicating more social support. Only the Social Interaction (4 items) and Subjective Social Support (7 items) subscales will be used.
Lubben social network scale - 6 (LSNS-6)- CHANGE IS BEING ASSESSED | Baseline, 4 month, 7 month
  The Lubben social network scale - 6 (LSNS-6) is a 6 item self-report measure of social engagement including family and friends. Scores range from 0-5 with higher scores indicating higher social engagement.
Patient-Reported Outcomes Measurement Information System (PROMIS) for Emotional Support and Informational Support- CHANGE IS BEING ASSESSED | Baseline, 4 month, 7 month
  The Patient-Reported Outcomes Measurement Information System (PROMIS) for Emotional Support and Informational Support consists of eight items each. The PROMIS Emotional Support (PROMIS-ES) measures the availability of others to speak with and feel appreciated by, whereas the PROMIS Informational Support (PROMIS-IS) measure captures perceived availability of advice or helpful information. Scores range from 1-5 with higher scores indicating higher support.
UCLA Loneliness Scale, Version 3 (UCLA)- CHANGE IS BEING ASSESSED | Baseline, 4 month, 7 month
  UCLA Loneliness Scale, Version 3 (UCLA) is a 20-item questionnaire that measures one's subjective feelings of loneliness and social isolation. Response options for each item range from 0 (Never) to 4 (often). Total scores range from 0 to 80 with higher scores indicating higher loneliness.
Interpersonal Needs Questionnaire-15 (INQ-15)- CHANGE IS BEING ASSESSED | Baseline, 4 month, 7 month
  The INQ-15 (19) is a self-report measure composed of 15 items that evaluate the main constructs of interpersonal suicide theory (8): PB (items 1-6), and TB (items 7-15). The items are answered on a 1-7 Likert scale with response options ranging from "Not at all true for me" to "Very true for me."
Client Satisfaction Questionaire-8 (CSQ-8)- CHANGE IS BEING ASSESSED | Baseline, 4 month, 7 month
  Client Satisfaction Questionaire-8 (CSQ-8) is an 8-item measure of participant satisfaction with the intervention. Scores on the CSQ-8 range from 8-32 with a higher score indicating higher satisfaction
VOICES Social Post-Interview (VSPI)- CHANGE IS BEING ASSESSED | Baseline, 4 month, 7 month
  VOICES Social Post-Interview (VSPI) is a brief interview (up to 30 minutes) that will consist of open and closed questions about initiation of the event, process of engaging with other participants, friend acquisition, as well as resources or key knowledge (e.g., healthcare, community opportunities) discovered.
Friend Acquisition Questionnaire- CHANGE IS BEING ASSESSED | Baseline, 4 month, 7 month
  Friend Acquisition Questionnaire is a 3-item questionnaire measuring utilization of the Veterans Socials for building structural social connections.
VS Facilitator Training Evaluation- CHANGE IS BEING ASSESSED | Baseline, 4 month
  The VS Facilitator Training Evaluation consists of approximately seventeen open and multiple-choice questions that immediately follow training and approximately four open and multiple-choice questions after a delay, when the VS facilitators begin implementing VS
VS Fidelity Checklist | Baseline, 4 month, 7 month-- CHANGE IS BEING ASSESSED
  The VS Fidelity Checklist measure consists of nineteen elements that guide facilitators through how best to maintain successful VS.
The Learning-Transfer Evaluation Model (LTEM)- CHANGE IS BEING ASSESSED | Baseline, 4 month, 7 month
  The Learning-Transfer Evaluation Model (LTEM) is an eight level model that divides the learning process into eight stages (attendance, activity, learner perceptions, knowledge, Decision making competence, task competence, transfer, and effects of transfer) and identifies the relevant assessment aspects for learning success at each stage.
The Berkman-Syme Social Network Index Adapted- CHANGE IS BEING ASSESSED | baseline. 4 month, 7 month
  a 4 item self report measure, and selected items will be used to assess the type, size, closeness, and frequency of contacts in a respondent's current social network. Respondents are categorized into four levels of social connection: socially isolated, moderately isolated, moderately integrated, and socially integrated. Scores range from 0 to 4, with 0 representing the highest level of social isolation and 4 representing the lowest level of social isolation.

CONTACTS AND LOCATIONS:
Overall Officials: Jay Gorman, PsyD, Principal Investigator — VA Bedford HealthCare System, Bedford, MA
Locations (1):
- VA Bedford HealthCare System, Bedford, MA, Bedford, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-02-27): https://cdn.clinicaltrials.gov/large-docs/34/NCT06145334/ICF_000.pdf